CLINICAL TRIAL: NCT06814509
Title: Delivering HOPE (Helping Women Optimize Prenatal Equity)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 298238
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Gestational Weight Gain; Diet, Healthy; Gestational Hypertension; Gestational Diabetes; Pregnancy Complications
MeSH Terms: conditions — Gestational Weight Gain; Hypertension, Pregnancy-Induced; Diabetes, Gestational; Pregnancy Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard of Care (ESoC) (Active Comparator): The ESoC arm includes implementing a standard clinical protocol for nutritional and gestational weight gain counseling recommended for all pregnant women; implementing a standard protocol for helping participants sign up for WIC and SNAP; and implementing a standard protocol for providing referrals to safety net food organizations.
  Interventions: Behavioral: Enhanced Standard of Care (ESoC)
- Delivering HOPE (Experimental): The Delivering HOPE arm includes providing the same nutritional and gestational weight gain counseling, WIC and SNAP assistance, and referral assistance as ESoC. In addition, participants in the Delivering HOPE arm will be provided with funds during their pregnancy to be used specifically for the purchase of healthy foods. The amount will vary based on household size as follows: $1,000 (one to two household members), $2,000 (three to four household members), or $3,000 (five plus household members).
  Interventions: Behavioral: Delivering HOPE

INTERVENTIONS:
Behavioral: Enhanced Standard of Care (ESoC) — Standard recommended nutrition and gestational weight gain counseling; WIC and SNAP enrollment assistance; emergency food referrals
  Arms: Enhanced Standard of Care (ESoC)
Behavioral: Delivering HOPE — ESoC plus healthy food provision
  Arms: Delivering HOPE

SUMMARY:
The overarching research question is: "Does the provision of healthy food (Delivering HOPE) during pregnancy reduce the proportion of women who experience excessive gestational weight gain compared with enhanced standard of care (ESoC)?" To answer this question, the investigators will conduct a large multi-site randomized controlled trial with 1,440 women. Women will be randomized to either the Delivering HOPE arm or the ESoC arm, with approximately 720 participants per arm. Participants randomized to the ESoC arm will receive the standard clinical protocol for nutritional and gestational weight gain counseling recommended for all pregnant women, WIC and SNAP enrollment assistance, referrals to safety net food organizations.Those randomized to the Delivering HOPE arm will be provided the same nutritional and gestational weight gain counseling, WIC and SNAP assistance, and food referrals, as well as a total of $1000/$2000/$3000 (depending on household size) during pregnancy to be used specifically for the purchase of healthy foods recommended in the nutritional counseling. Data for the primary outcome (pre-pregnancy weight and weight at delivery) will be collected from birth records.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-44 years
* ≤18 weeks pregnant
* Speak English, Spanish, or Marshallese
* Valid email address

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1440 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Excessive gestational weight gain (EGWG) | Baseline to Post-partum (approx. 40 weeks)
  Pre-pregnancy weight and weight immediately prior to birth will be used to calculate total weight gain, adjusting for pre-pregnancy body mass index and weeks of gestation. Individuals whose total weight gain exceeds established guidelines will be determined to have EGWG. We will examine the difference in the proportion of women who experience EGWG.

CONTACTS AND LOCATIONS:
Overall Officials: Pearl McElfish, PhD, Principal Investigator — University of Arkansas; Lanita White, PharmD, Principal Investigator — Community Health Centers of Arkansas
Locations (8):
- United States (8):
  - 1st Choice Healthcare, Corning, Arkansas
  - River Valley Primary Care Services, Lavaca, Arkansas
  - Olly Neal Community Health Center, Marianna, Arkansas
  - Boston Mountain Rural Health Center, Marshall, Arkansas
  - Mainline Health Systems, Monticello, Arkansas
  - Jefferson Comprehensive Care System, Pine Bluff, Arkansas
  - Community Clinic, Springdale, Arkansas
  - East Arkansas Family Health Center, West Memphis, Arkansas

IPD SHARING:
Plan to Share IPD: No